CLINICAL TRIAL: NCT00127569
Title: Multicenter, Phase II Trial Assessing the Efficacy of Rituximab in HIV Infected Patients With Multicentric Castleman Disease Dependent on Chemotherapy (ANRS 117 Study, CastlemaB)
Brief Title: Rituximab in the Treatment of HIV Associated Multicentric Castleman Disease Dependent on Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 117 CastlemaB
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2007-01-12 (Estimated); Status verified 2007-01

CONDITIONS: HIV Infections; Giant Lymph Node Hyperplasia
Keywords: HIV infections; Giant Lymph Node Hyperplasia; Herpesvirus 8, Human; Rituximab (Mabthera); Antibodies, Monoclonal
MeSH Terms: conditions — HIV Infections; Castleman Disease; Sarcoma, Kaposi | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This trial is aimed to study the efficacy of 4 weekly cycles of rituximab in HIV-infected patients with multicentric Castleman disease (giant lymph node hyperplasia) dependent on chemotherapy. Efficacy is assessed by the complete response rate at day 60. The patients are followed until day 365.

DETAILED DESCRIPTION:
HIV-related multicentric Castleman disease (MCD) is a lymphoproliferative disorder characterized by lymphadenopathy with angiofollicular hyperplasia and plasma cell infiltration, associated with KSHV/HHV-8. Patients typically have systemic manifestations such as fever associated with lymphadenopathy, hepatosplenomegaly, respiratory symptoms, peripheral edema, cytopenia, hypergammaglobulinemia, hypoalbuminemia, and high levels of serum C reactive protein (CRP). Symptoms correlate with an important increase of KSHV/HHV-8 DNA in peripheral blood mononuclear cells. HIV-MCD is characterized by a rapidly progressive and often fatal course. HIV-MCD is often refractory to treatment. Vinca alkaloids produce frequent but short-lived responses, and most patients remain dependant upon chemotherapy.

Lymph nodes of patients with HIV-MCD specifically harbor the virus in B cells located in the mantle zone, which stain positively for the CD20 surface antigen. Rituximab, a humanized monoclonal anti-CD20 antibody, has been reported to be effective in some cases, with conflicting data in other cases. The optimal schedule of infusions remains unclear.

Kaposi's sarcoma is often associated with HIV-MCD, and the development of aggressive non-Hodgkin's lymphoma is not a rare outcome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed multicentric Castleman disease, with dependence on vinblastine or VP16 for at least 3 months, whenever they have been splenectomized
* At least one Castleman crisis since onset of chemotherapy
* Ongoing highly active antiretroviral therapy (HAART) for at least 3 months
* No threshold of CD4 cell count and HIV-RNA
* Signed written informed consent

Exclusion Criteria:

* Prior treatment with rituximab
* Evolutive lymphoma or Kaposi's sarcoma needing treatment
* Absence of effective contraception
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-05; Study Completion 2006-01

PRIMARY OUTCOMES:
Sustained response rate of multicentric Castleman disease at day 60, after 4 infusions of rituximab

SECONDARY OUTCOMES:
One-year disease-free survival
One-year event-free survival
Relapse rate at day 365
One-year lymphoma-free survival
Tolerance of rituximab
One-year overall survival
Change in HHV-8 viral load within one year
Change in lymphocyte B cell count within one year

CONTACTS AND LOCATIONS:
Overall Officials: Eric Oksenhendler, M.D., Principal Investigator — AP-HP Hopital Saint-Louis